CLINICAL TRIAL: NCT00095550
Title: The Efficacy and Safety of Irbesartan/HCTZ Combination Therapy as First Line Treatment for Patients With Moderate Hypertension
Brief Title: Irbesartan/Hydrochlorothiazide (HCTZ) Combination Therapy for Patients With Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-185
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: Moderate Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A1 (Experimental)
  Interventions: Drug: Irbesartan/HCTZ
- A2 (Active Comparator)
  Interventions: Drug: Irbesartan monotherapy
- A3 (Active Comparator)
  Interventions: Drug: HCTZ monotherapy

INTERVENTIONS:
Drug: Irbesartan/HCTZ — Tablets, Oral, Irbesartan 150 mg/HCTZ 12.5 mg, Once daily, 12 weeks.
  Other Names: Avapro
  Arms: A1
Drug: Irbesartan monotherapy — Tablets, Oral, 150 mg, Once daily, 12 weeks.
  Other Names: Avapro
  Arms: A2
Drug: HCTZ monotherapy — Tablets, Oral, 12.5 mg, Once daily, 12 weeks.
  Arms: A3

SUMMARY:
The purpose of this clinical research is to learn if moderate hypertension can be better controlled by initially treating with a combination of drugs (Irbesartan/HCTZ), in patients who are unlikely to achieve blood pressure (B/P) control with only one drug. In addition, the study will also evaluate the safety and tolerability of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Subjects must have uncontrolled hypertension defined as:

  * average systolic blood pressure between 160 mmHg and 180 mmHg (while diastolic blood pressure is less than 110 mmHg) or
  * average diastolic blood pressure between 100 mmHg and 110 mmHg (while systolic blood pressure is between 130 mmHg and 180 mmHg)
* Subjects must be willing to discontinue their antihypertensive medication, if applicable.
* Men and women, ages 18 and older will be included.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to one week after the study in such a manner that the risk of pregnancy is minimized. WOCBP must have a negative serum or urine pregnancy test within 72 hours prior to the start of study medication.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Known or suspected secondary hypertension
* Hypertension emergencies or stroke within the past 12 months.
* Heart attack, angina or bypass surgery within the past six months.
* Significant kidney disease
* Significant liver disease
* Systemic lupus erythematosus
* Gastrointestinal disease or surgery that interfere with drug absorption
* Cancer during the past five years excluding localized squamous cell or basal cell carcinoma of the skin
* Currently pregnant or lactating
* Mental condition (psychiatric or organic cerebral disease) rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Drug or alcohol abuse within the last five years
* Known allergy to irbesartan or diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in SeSBP at Week 8

SECONDARY OUTCOMES:
Frequency of discontinuation due to AE, frequencies of hypotension, dizziness, syncope, headaches, hypokalemia and hyperkalemia after 12 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (128):
- United States (87):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Columbiana, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Carmichael, California
  - Local Institution, Fair Oaks, California
  - Local Institution, Fresno, California
  - Local Institution, Long Beach, California
  - Local Institution, Rolling Hills Estate, California
  - Local Institution, Roseville, California
  - Local Institution, Sacramento, California
  - Local Institution, San Jose, California
  - Local Institution, Torrance, California
  - Local Institution, Tustin, California
  - Local Institution, Highlands Ranch, Colorado
  - Local Institution, Bridgeport, Connecticut
  - Local Institution, Waterbury, Connecticut
  - Local Institution, Newark, Delaware
  - Local Institution, Chipley, Florida
  - Local Institution, Clearwater, Florida
  - Local Institution, Crestview, Florida
  - Local Institution, DeLand, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Niceville, Florida
  - Local Institution, Ocoee, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Saint Cloud, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Peoria, Illinois
  - Local Institution, Chalmette, Louisiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Oxon Hill, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Livonia, Michigan
  - Local Institution, Saginaw, Michigan
  - Local Institution, Olive Branch, Mississippi
  - Local Institution, Missoula, Montana
  - Local Institution, Dover, New Hampshire
  - Local Institution, South Bound Brook, New Jersey
  - Local Institution, Buffalo, New York
  - Local Institution, Mount Vernon, New York
  - Local Institution, New York, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Gastonia, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Mint Hill, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Canton, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Genoa, Ohio
  - Local Institution, Kettering, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Medford, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Bensalem, Pennsylvania
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution, Collegeville, Pennsylvania
  - Local Institution, Levittown, Pennsylvania
  - Local Institution, Penndel, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, West Grove, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Columbia, South Carolina
  - Local Institution, Orangeburg, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Summerville, South Carolina
  - Local Institution, Bartlett, Tennessee
  - Local Institution, Hendersonville, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Selmer, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Colleyville, Texas
  - Local Institution, Midland, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Olympia, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Madison, Wisconsin
  - Local Institution, Milwaukee, Wisconsin
- Canada (22):
  - Local Institution, Red Deer, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, North Vancouver, British Columbia
  - Local Institution, Sidney, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Aylmer, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Markham, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Richmond Hill, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montague, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- France (4):
  - Local Institution, Angers
  - Local Institution, Bouchemaine
  - Local Institution, Briollay
  - Local Institution, Tiercé
- Germany (12):
  - Local Institution, Spaichingen, Baden-Wurttembe
  - Local Institution, Spaichingen, Braden-Wurttembe
  - Local Institution, Berlin
  - Local Institution, Essen
  - Local Institution, Feldafing
  - Local Institution, Grömitz
  - Local Institution, Künzing
  - Local Institution, Nörten-Hardenberg
  - Local Institution, Nuremberg
  - Local Institution, Ornbau
  - Local Institution, Unterschneidheim
  - Local Institution, Villingen-Schwenningen
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov